CLINICAL TRIAL: NCT02181777
Title: Exploring the Feasibility of Social Skills Training in People With Psychosis.
Brief Title: Group Training for Social Skills in Psychosis
Acronym: GRASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Matteo Cella, Principal Investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R&D2014/018
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Psychotic Disorders
Keywords: Psychosis; Schizophrenia; Social Skills; Therapy
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Social Skills | interventions — Hand Strength; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GRASP (Experimental): GRoup trAining for Social skills in Psychosis
  Interventions: Behavioral: GRASP
- Standard care (Active Comparator): Treatment as usual as provided by care team
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: GRASP — GRoup trAining for Social skills in Psychosis
  Arms: GRASP
Behavioral: Standard care — Treatment as usual
  Arms: Standard care

SUMMARY:
The purpose of this study is to assess the feasibility of a social skills training group for people with psychosis.

DETAILED DESCRIPTION:
This study is assessing the feasibility of a psychological intervention targeting social cognition problems in people with psychosis. The intervention is a group psychological treatment facilitated by a clinical psychologist. The group therapy takes advantage of audiovisual material and practical exercises to illustrate strategies and thinking styles that may help participants overcome difficulties in social settings.

A second objective of this study is to test a new method to measure social cognition by using portable devices. These devices will be carried by participants in their everyday life and will ask about their social activity levels at random times and record activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis part of the psychosis spectrum (according to DSM-IV or DSM-V or ICD-10)
* Good command of the English language
* Social engagement problems as evidenced by care coordinator report and number of hours spent in social activities per week lower than 10.

Exclusion Criteria:

* Primary diagnosis of substance abuse disorder
* Change in antipsychotic medication in the last six weeks
* Significant learning difficulties (premorbid IQ lower than 70)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12-31 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Therapy drop-out rate | 8 weeks post randomisation
Number of therapy session attended | 8 weeks post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Cella, DClinPsy, Principal Investigator — Institute of Psychiatry
Locations (1):
- Kings College London, London, United Kingdom

REFERENCES:
- [Background] Penn DL, Roberts DL, Combs D, Sterne A. Best practices: The development of the Social Cognition and Interaction Training program for schizophrenia spectrum disorders. Psychiatr Serv. 2007 Apr;58(4):449-51. doi: 10.1176/ps.2007.58.4.449. PMID 17412842
- See also: Related Information — https://www.ukcrc.org/research-infrastructure/clinical-research-networks/uk-clinical-research-network-ukcrn/